CLINICAL TRIAL: NCT06894147
Title: "Comparison of the Effects of Genicular Radiofrequency Ablation and Pulsed Radiofrequency Applications on Pain Levels in Patients with Osteoarthritis, Guided by Ultrasound''
Brief Title: Genicular Radiofrequency Ablation Versus Pulsed Radiofrequency
Acronym: GRFT-PRF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ülkü Sabuncu, Assoc. Prof., Ankara City Hospital Bilkent
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: TABED-1-24-88
Record Dates: First submitted 2025-03-07; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis of Knee
Keywords: Osteoarthritis of Knee; Pulsed Radio Frequency Treatment; Radiofrequency Ablation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized Controlled, Double-Blind
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient Blinding (Single Blind for Patients):
  The patients will not be informed about which treatment group they have been assigned to.
  They will only know that they are participating in a clinical trial, but not the specifics of the treatment or control group.
  Investigator Blinding (Double Blind for Investigators):
  The principal investigator and all clinical staff involved in the treatment administration and assessment of outcomes will also be blinded to the patients' group assignments.
  The study medications or interventions will be labeled with codes, and the investigators will not have access to the key linking these codes to the specific treatments.
  Randomization:
  Random assignment will be used to allocate participants to one of the two groups (treatment group or control group) to ensure unbiased distribution of participants.
  Randomization will be performed using a computerized random number generator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiofrequency ablation (Experimental): After performing a diagnostic block with 1 mL of 1% lidocaine on the superior medial, lateral, and inferior medial genicular nerve branches, patients who experience more than 50% benefit from the procedure will undergo radiofrequency ablation on the genicular nerve branches.
  Interventions: Procedure: Genicular nerve pulse radiofrequency
- Pulsed radiofrequency (Experimental): After performing a diagnostic block with 1 mL of 1% lidocaine on the superior medial, lateral, and inferior medial genicular nerve branches, patients who experience more than 50% benefit from the procedure will undergo either pulsed radiofrequency on the genicular nerve branches.
  Interventions: Procedure: Genicular nerve pulse radiofrequency

INTERVENTIONS:
Procedure: Genicular nerve pulse radiofrequency — After performing a diagnostic block with 1 mL of 1% lidocaine on the superior medial, lateral, and inferior medial genicular nerve branches, patients who experience more than 50% benefit from the procedure will undergo pulsed radiofrequency aplication.

SUMMARY:
This study investigates the effectiveness of two treatments-genicular nerve radiofrequency ablation and pulsed radiofrequency-in reducing pain and improving function in osteoarthritis patients. These techniques, used after diagnostic nerve blocks, aim to provide long-lasting pain relief. Despite both being found effective, no clear consensus exists on which method is superior. The study seeks to compare these techniques and contribute new insights to the existing literature.

DETAILED DESCRIPTION:
Chronic knee pain, especially in osteoarthritis patients, is a common condition that significantly affects mobility and quality of life. In individuals over the age of 60, the incidence is 9.6% in men and 18% in women. In patients with osteoarthritis, weight loss and appropriate exercises are recommended as the primary treatments. This is followed by medical therapy, injection treatments, and, if necessary, total knee arthroplasty. However, for patients with a body mass index (BMI) of 40 or higher, total knee arthroplasty is avoided due to the high surgical risk. In recent years, genicular nerve diagnostic block and radiofrequency ablation have been shown to reduce pain and improve function in these patients . Radiofrequency ablation works by blocking the transmission of sensory nerves, thereby improving function.

The innervation of the knee joint originates from the femoral nerve's articular branches, the common peroneal, saphenous, tibial, and obturator nerves. These articular branches are known as the genicular nerves, which are superficial and can be easily accessed using both fluoroscopy and ultrasound.

In osteoarthritis patients, superior medial, superior lateral, and inferior medial genicular nerve blocks are applied. After the diagnostic block, some clinics apply radiofrequency thermocoagulation to the genicular nerve branches for a lasting effect, while others use pulsed radiofrequency. Both techniques have been found to be effective, but there is no data in the literature regarding which technique is superior. The aim of this study is to determine which of the two techniques is more effective and share the findings with the literature.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18
* osteoarthritis
* Grade 2-4 gonarthrosis according to the Kellgren-Lawrence (KL) classification
* Pain 6-10 on the Numeric Rating Scale (NRS)

Exclusion Criteria:

* Patients with chronic knee pain due to another pathology (e.g., meniscopathy, trauma, rheumatoid arthritis) History of previous knee surgery History of intra-articular injection in the last 3 months Coagulopathy, use of antiplatelet or anticoagulant medications Infection Severe psychiatric disorders Patients with a cardiac pacemaker or defibrillator Renal or hepatic failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) , | Baseline, 3 weeks, 3 months.
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable

SECONDARY OUTCOMES:
Western Ontario and McMaster (WOMAC) Osteoarthritis Index | Baseline, 3 weeks, 3 months.
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
privacy.

REFERENCES:
- [Background] Kirdemir P, Catav S, Alkaya Solmaz F. The genicular nerve: radiofrequency lesion application for chronic knee pain. Turk J Med Sci. 2017 Feb 27;47(1):268-272. doi: 10.3906/sag-1601-171. PMID 28263500
- [Background] Fitzpatrick B, Cowling M, Poliak-Tunis M, Miller K. Effect of Genicular Nerve Radiofrequency Ablation for Knee Osteoarthritis: A Retrospective Chart Review. WMJ. 2021 Jul;120(2):156-159. PMID 34255959